CLINICAL TRIAL: NCT01126307
Title: Study of Verapamil in Refractory Epilepsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Dr. Danielle Andrade, Toronto Western Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UHN REB # 10-0024-A
Record Dates: First submitted 2010-05-17; First posted 2010-05-19 (Estimated); Last update posted 2010-05-19 (Estimated); Status verified 2010-03

CONDITIONS: Epilepsy; Seizures
Keywords: refractory epilepsy- greater than 4 seizures in 2 month baseline period
MeSH Terms: conditions — Epilepsy; Seizures | interventions — Verapamil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- verapamil (Active Comparator): verapamil 80mg tid
  Interventions: Drug: Verapamil
- placebo sugar pill (Placebo Comparator): placebo tid
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Verapamil — 80 mg tid
  Other Names: Isoptin
  Arms: verapamil
Drug: placebo — placebo tid
  Arms: placebo sugar pill

SUMMARY:
Epilepsy is one of the most common chronic neurological diseases, affecting 300,000 Canadians. One in 3 epilepsy patients have refractory seizures meaning that all antiseizure drugs fail to control their seizures. This drug resistance in epilepsy may be related to the over expression of multidrug resistance proteins (MDR). Varapamil inhibits MDR. We propose to add verapamil/placebo to patients' anti epilepsy medication for 3 months. Patients who receive placebo will have verapamil added for 3 months after the completion of the double-blind treatment period. Seizure frequency/severity will be tracked. Blood samples for DNA will be collected. There will be 9 clinic visits over 32 weeks. ECG and echocardiogram will be done at baseline and repeated if necessary

DETAILED DESCRIPTION:
This open label study will consist of three phases: baseline, Double-blind treatment and open-label-treatment. There are 9 visits over 32 weeks. During the baseline period, the number of seizures will be recorded during 2 months while the patient is on a dose of antiseizure drug(s) that was previously established to provide better seizure control. Blood work, including blood for DNA baseline ECG and echocardiogram will be done and may be repeated if necessary. During the 3 months of double-blind treatment phase, verapamil/placebo will be added to the current medications. Visits are every 4 weeks. Vital signs, seizure counts and adverse events will be evaluated. All patients who received placebo will be offered 3 months of open-label treatment with verapamil.

ELIGIBILITY:
Inclusion Criteria:

* 1. patients in whom seizures are not controlled by their antiseizure medication;
* 2. must have at least 2 seizures per month.

Exclusion Criteria:

* Exclusion: patients with cardiovascular problems that could be adversely affected by verapamil

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2010-06; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
percentage reduction of seizure frequency | 3 months
  after 3 months of treartment compared to baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada